CLINICAL TRIAL: NCT05968235
Title: Association of Glucose and Lipid Metabolism Levels and Vitiligo : a Case-control Study
Brief Title: Correlation of Glucose and Lipid Metabolism Levels With Vitiligo
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Li Chunying-1, Vice Chief, Xijing Hospital
Other Study IDs: XJPF-LCY-V202307
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Metabolism Disorder, Glucose; Metabolism Disorder, Lipid; Vitiligo
Keywords: Vitiligo; Glucose; Lipid
MeSH Terms: conditions — Glucose Metabolism Disorders; Lipid Metabolism Disorders; Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples of vitiligo patients and healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitiligo: Patients diagnosed with vitiligo
  Interventions: Other: Collecting blood samples
- Healthy: Healthy volunteers with sex- and age-matched with vitiligo patients
  Interventions: Other: Collecting blood samples

INTERVENTIONS:
Other: Collecting blood samples — Peripheral blood was collected from the study subjects and blood glucose, glycosylated hemoglobin, triglycerides, total cholesterol, high-density lipoprotein and low-density lipoprotein levels were measured in the peripheral blood.

SUMMARY:
The goal of this observational study is to compare serum glucose and lipid metabolism levels between health volunteers and vitiligo patients. The main question it aims to answer is whether vitiligo is related to glucose and lipid metabolism disorders. Participants will complete a vitiligo questionnaire and test serum levels of indicators related to glucose and lipid metabolism. Researchers will compare vitiligo patients with healthy volunteers to see if there is a correlation between vitiligo and disorders of glucose and lipid metabolism.

DETAILED DESCRIPTION:
Vitiligo is a common autoimmune skin disease, which causes white spot formation due to destruction of epidermal melanocytes, severely affecting the physical and mental health of patients, but treatment is extremely difficult due to unclear pathogenesis. Studies have reported that patients with type I diabetes mellitus combined with vitiligo, the risk of metabolic syndrome, diabetes mellitus, elevated lipids, and obesity in vitiligo patients is higher than that of healthy controls, and other studies have reported that vitiligo lesions in patients with hypercholesterolemia combined with vitiligo treated with simvastatin get rapid skin color, suggesting that there is a correlation between glucose and lipid metabolism and the vitiligo disease, but as of now there is no research study on the correlation of glucose and lipid metabolism and vitiligo pathogenesis, much less large data can be analyzed for reference. Therefore, there is an urgent need to study the metabolic profile of vitiligo patients and utilize the basic research platform to explore the role of abnormal body metabolism in the onset or progression of vitiligo.

This study intends to conduct a cross-sectional study, using questionnaires to collect and register vitiligo patients' disease information, etc., to establish a database of study subjects, and to collect peripheral blood samples from vitiligo patients to test the levels of key indicators of glycolipid and lipid metabolism, and to analyze their correlation with clinical features, disease activity, and treatment of vitiligo. Through the above studies, clinical evidence for the involvement of abnormalities in glycolipid and lipid metabolism in the development of vitiligo was provided.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as vitiligo by a dermatologist based on a combination of clinical manifestations (milky white or porcelain white patches), Wood's Lamp test results (bright white fluorescence), and histopathologic test results (reduction or disappearance of epidermal melanocytes in the white patches);
2. Male or female subjects, age between 18 and 60 years old;
3. Stable vital signs;
4. Study subjects voluntarily signed an informed consent form.

Exclusion Criteria:

1. Subjects who have been systematically using glucocorticoids, immunosuppressants, etc. that affect glycolipid levels due to a combination of diseases other than metabolic diseases in the last 3 months shall be asked and determined by a clinician;
2. Women who are pregnant or breastfeeding shall be asked and determined by a clinician;
3. Subjects who suffer from psychiatric disorders, etc. and who are not capable of cooperating with the follow-up study shall be asked and determined by a clinician.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We recruited patients with clinically diagnosed vitiligo and age- and sex-matched healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Demographic and epidemiological information of the study subjects | 2020.02.01-2023.03.25
  Detailed records of demographic information (age, gender, occupation, education degree, life history, et al.), clinical information of vitiligo (age at onset, duration, severity, type, treatment, complication, et al.) and physical examination index (height, weight, blood pressure, heart rate).
Serum glucose and lipid metabolism levels of the study subjects | 2020.02.01-2023.03.25
  Detection of fasting blood glucose, glycosylated hemoglobin, triglycerides, total cholesterol, high-density lipoproteins, and low-density lipoproteins in peripheral blood of study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chunying Li, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided